CLINICAL TRIAL: NCT05894265
Title: Prospective Pilot Study to Determine the Safety and Effectiveness of a Connective Tissue Allograft (Active Matrix) vs. Standard of Care in Arthroscopic Rotator Cuff Repair
Brief Title: Prospective Study to Determine the Safety and Effectiveness of a Connective Tissue Allograft Active Matrix (AM) vs. Standard of Care in Arthroscopic Rotator Cuff Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Skye Biologics Holdings, LLC (Industry)
Responsible Party: Principal Investigator, Eric F Berkman, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-23-0312
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Rotator Cuff Tears
Keywords: musculoskeletal injuries; rotator cuff repair
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ActiveMatrix® Dosage A (Experimental)
  Interventions: Other: ActiveMatrix® Dosage A
- ActiveMatrix® Dosage B (Experimental)
  Interventions: Other: ActiveMatrix® Dosage B
- Saline Injection (Placebo Comparator)
  Interventions: Procedure: Saline injection

INTERVENTIONS:
Other: ActiveMatrix® Dosage A — This group will receive ActiveMatrix® (AM) product dosage A (1cc AM diluted to 3cc with saline)
  Other Names: Human Placental Connective Tissue-Derived Allograft
  Arms: ActiveMatrix® Dosage A
Other: ActiveMatrix® Dosage B — Group 2 will receive ActiveMatrix® product dosage B (2cc AM diluted to 3cc with saline)
  Other Names: Human Placental Connective Tissue-Derived Allograft
  Arms: ActiveMatrix® Dosage B
Procedure: Saline injection — Group 3 will receive saline injection
  Arms: Saline Injection

SUMMARY:
The purpose of this study is to see how well the ActiveMatrix® graft works at improving healing and function of the shoulder following rotator cuff repair surgery

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* 1-2 tendon full thickness reparable rotator cuff tendon tear(s)

Reparable tear defined as:

a tear of the rotator cuff where it is possible to bring the retracted tendon edge back to the greater tuberosity of the humerus under minimal tension.

Full-thickness tear defined as:

a tear that involves the majority of supraspinatus and less than half of the infraspinatus under minimal tension, with no subscapularis involvement beyond the upper border

* Failed conservative medical management of the rotator cuff tendon tear defined as: 4-6 weeks of formal physical therapy or guided home exercises and activity modification
* Have no contraindications or allergies to the treatment administered
* Have current imaging studies (plain radiographs and MRI exams) of the shoulder to rule out other etiologic diagnoses
* Able and willing to comply with the post-operative physical therapy and study follow-up schedule

Exclusion Criteria:

* Prior surgery on the index shoulder within 12 months of enrollment, including Latarjet procedures, superior labral treat from anterior to posterior (SLAP), and (failed) primary rotator cuff surgery,
* Prior surgery for bone defects requiring bone implantation in the index shoulder,
* Steroid injection into the index shoulder within 6 weeks of enrollment.
* Subscapularis tear greater than 1/3 of tendon involvement requiring repair,
* Calcific tendonitis in the index shoulder,
* Fatty infiltration of the index shoulder rotator cuff muscle, i.e. Goutallier classification ≥ Grade 3,
* Contralateral shoulder injury that may interfere with the post-operative rotator cuff repair rehab guidelines,
* History of advanced osteoarthritis of glenohumeral joint (AC joint can have advanced OA) i.e. Samilson-Prieto classification ≥ Grade 2
* History of malignant tumor and osseous metastatic disease,
* History of heterotopic ossification,
* History of chronic pain disorders (i.e., fibromyalgia),
* Current substance abuse (drug or alcohol), by the investigator's judgment,
* For females of child-bearing potential: unable or unwilling to take adequate contraceptive precautions during the study, known to be pregnant at enrollment, breastfeeding an infant at enrollment or during the study, or planning to become pregnant during the study,
* Currently participating in, or have been recently exited from (within 30 days from enrollment in this study), or plan to enroll in another clinical study for a bone allograft or drug that may impact participation or outcomes of this study,
* Currently involved in any injury litigation or workers compensation claims,
* has a condition, disorder or other factor that, in the investigator's opinion, would interfere with study participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Sugaya score as measured by Magnetic Resonance Imaging (MRI) | 6 months post surgery , 12 months post surgery
  Sugaya classification is a classification system that is used to analyze postoperative rotator cuff tendon integrity

SECONDARY OUTCOMES:
Change in range of motion as assessed by the Passive Range of Motion (PROM) assessment using a goniometer | baseline, 4weeks, 3 months, 6 months 9 months, and 12 months
  A goniometer will be used to measure range of motion during the PROM assessment. The goniometer measures the angle between the beginning position and the ending position of available motion, and the result is reported in degrees.PROM will be measured on both sides
Change in shoulder function as assessed by the American Shoulder and Elbow Surgeons Shoulder Score (ASES) | baseline, 4weeks, 3 months, 6 months 9 months, and 12 months
  The total score is weighted 50% for pain and 50% for function. The pain score is calculated by subtracting the VAS from 10 and multiplying it by 5. The 10 functional questions are scored on a 4-point scale (0-3) with a maximum functional score of 30. The raw functional score is then multiplied by 5/3 to make the maximum functional score out of 50 possible points. The pain and function scores are then added together to obtain the final ASES score (out of 100). Higher scores correlate to better outcomes.
Change in pain intensity as assessed by the Visual Analog Scale (VAS) | baseline, 4weeks, 3 months, 6 months 9 months, and 12 months
  VAS is scored on a 100mm horizontal scale that represents the patients pain intensity. A higher score corresponds to increased pain intensity
Change in pain and functional disability as assessed by the Shoulder Pain and Disability Index (SPADI) | baseline, 4weeks, 3 months, 6 months 9 months, and 12 months
  SPADI is a self-administered questionnaire that measures a combination of pain and functional disability. This contains 13 items that assess two domains; a 5-item subscale that measures pain and an 8-item subscale that measures disability and each is scored from 0 = no pain and 10 = the worst pain imaginable. SPADI is scored from 0 to 130 with a high score representing more pain and disability.

CONTACTS AND LOCATIONS:
Overall Officials: Eric F Berkman, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No